CLINICAL TRIAL: NCT04392414
Title: Randomized, Open Label, Prospective Study of the Safety and Efficacy of Hyperimmune Convalescent Plasma in Moderate and Severe COVID-19 Disease
Brief Title: Hyperimmune Convalescent Plasma in Moderate and Severe COVID-19 Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CovPlas-Covid19
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 convalescent hyperimmune plasma (Experimental): Moderately and severely ill COVID-19 patients treated with convalescent hyperimmune plasma. Patients will be infused with two units of 300 ml
  Interventions: Biological: COVID-19 convalescent hyperimmune plasma
- Non-convalescent fresh frozen plasma (Standard plasma) (Placebo Comparator): Moderately and severely ill COVID-19 patients treated with non-convalescent fresh frozen plasma (standard plasma). Patients will be infused with two units of 300 ml
  Interventions: Biological: Non-convalescent fresh frozen plasma (Standard plasma)

INTERVENTIONS:
Biological: COVID-19 convalescent hyperimmune plasma — Subjects to receive double convalescent hyperimmune plasma units of 300 ml each, with the 2nd unit administered no later than 24 hrs after the first one
  Arms: COVID-19 convalescent hyperimmune plasma
Biological: Non-convalescent fresh frozen plasma (Standard plasma) — Subjects to receive double standard plasma units of 300 ml each, with the 2nd unit administered no later than 24 hrs after the first one
  Arms: Non-convalescent fresh frozen plasma (Standard plasma)

SUMMARY:
The clinical trial aims to study the safety and efficacy of transfusion of COVID-19 convalescent hyperimmune plasma for the treatment of moderate and severe forms of COVID-19 disease in comparison with non-convalescent fresh frozen plasma (standard plasma).

DETAILED DESCRIPTION:
This is a study of the safety and efficacy of the use of COVID-19 convalescent plasma (from subjects who have recovered from SARS-CoV-2) in the treatment of moderate and severe forms of the SARS-CoV-2 infection. Currently, there are no registered drugs for the treatment of the SARS-CoV-2 infection in the world. The use of hyperimmune plasma is a well-known method used for many decades to treat many dangerous infections. The effectiveness of such a therapy for COVID-19 patients has recently been demonstrated in a number of clinical studies in China. Therefore, we plan to study the feasibility of administering multiple doses of COVID-19 convalescent plasma in comparison with standard plasma to moderate and severe patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-75 years.
2. The presence of COVID-19 infection, confirmed by PCR testing
3. The presence of the COVID-19 pneumonia pattern on the chest HRCT with a damage to more than 25% of the lung parenchyma
4. Morning fever ≥ 38.0 °C over the last three days
5. CRP blood level ≥ 50 mg / ml or ferritin blood level ≥ 600 μg / ml
6. A signed informed consent

Exclusion Criteria:

1. Respiratory index ≤200
2. Contraindications for the transfusion of donor immune plasma or history of prior reactions to blood transfusions
3. Mechanical ventilation
4. The presence of chronic lung diseases with chronic respiratory failure.
5. The need for home continuous oxygen therapy before the onset of current disease.
6. Serum creatinine level higher than 150 μmol / l
7. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
The number and proportion of patients with the normal body temperature (≤37.2 C) at the day 1, 2, 3, 4, 5, 6, 7 after the start of therapy | Days 1, 2, 3, 4, 5, 6, 7
  The number and proportion of patients with the normal body temperature (≤37.2 C) at the days 1, 2, 3, 4, 5, 6, 7 after the start of therapy, for the statistical data comparison between the two arms.

SECONDARY OUTCOMES:
Days before mechanical ventilation | 30 days
  For each patient, the number of days passed from the plasma administration to placing on mechanical ventilation will be noted, for the statistical data comparison between the two arms.
Days of need for oxygen therapy | 30 days
  For each patient, the number of days he or she spent on the oxygen support after the plasma administration will be noted, for the statistical data comparison between the two arms.
Days of stay in the ICU | 30 days
  For each patient, the entire duration of ICU stay after the plasma administration will be noted, for the statistical data comparison between the two arms.
Days of hospitalization | 30 days
  For each patient, the entire duration of hospital stay after the plasma administration will be noted, for the statistical data comparison between the two arms.
Changes of the titer of the SARS-CoV-2 antibodies in the blood plasma of patients | Days 0, 14, 30
  Changes of the plasma levels of the SARS-CoV-2 antibodies, days 14 and 30 after the treatment start vs those levels before the treatment start (day 0) for the same patients.
Dynamics of the cytokine profile | Days 0, 3, 7
  Changes of the plasma levels of IL2, IL6, IL10, TNFalpha and INFgamma, days 3 and 7 after the treatment start vs those levels before the treatment start (day 0) for the same patients.
Incidence of the cytokine storm development and the need of administering cytokine storm inhibitors | Days 3, 7
  Incidence of administering IL6 receptor blockers (tocilizumab, sarilumab)
Dynamics of the level of C-reactive protein | Days 0, 1, 2, 3, 4, 5, 6, 7
  Changes of the plasma levels of C-reactive protein, days 1, 2, 3, 4, 5, 6, 7 after the treatment start vs those levels before the treatment start (Day 0) for the same patients.
30-day mortality rate | 30 days
  30-day mortality rate, for the statistical data comparison between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Averyanov, MD, PhD, Principal Investigator — Federal Pulmonology Scientific and Research Institute, FMBA of Russia; Vladimir P Baklaushev, MD, PhD, Study Director — Federal Research Clinical Center, FMBA of Russia
Locations (1):
- Federal Research Clinical Center of Federal Medical & Biological Agency, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD).

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969